CLINICAL TRIAL: NCT06317558
Title: Real-world Clinical Outcomes of Neoadjuvant Immunotherapy in NSCLC Patients: A Retrospective, Multi-center, Cohort Study (NeoIM-Lung)
Brief Title: Real-world Clinical Outcomes of NSCLC Patients Receiving Neoadjuvant Immunotherapy
Acronym: NeoIM-Lung
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 22/492-3694
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: NSCLC
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Neoadjuvant immunotherapy: Immune checkpoint inhibitors are used for neoadjuvant treatment in this cohort.
  Interventions: Drug: Neoadjuvant immunotherapy
- Other neoadjuvant treatment: Other drugs other than Immune checkpoint inhibitors are used for neoadjuvant treatment in this cohort.
  Interventions: Drug: Other drugs for neoadjuvant treatment

INTERVENTIONS:
Drug: Neoadjuvant immunotherapy — Immune checkpoint inhibitors are used as neoadjuvant settings for NSCLC patients.
  Other Names: Immune checkpoint inhibitors
  Groups: Neoadjuvant immunotherapy
Drug: Other drugs for neoadjuvant treatment — Drugs other than immune checkpoint inhibitors are being used as a new adjuvant setting for patients with NSCLC.
  Other Names: Other drugs
  Groups: Other neoadjuvant treatment

SUMMARY:
The goal of this observational study is to evaluate the efficacy and long-term clinical outcomes of different neoadjuvant immunotherapies in non-small cell lung cancer (NSCLC) patients using the real-world data. The main questions it aims to answer are:

* What the best setting for immune checkpoint inhibitors as the neoadjuvant treatment?
* How to determine the subgroups of patients benefit from neoadjuvant immunotherapy? Participants will receive neoadjuvant immunotherapy the study will analyze the real-world data.

DETAILED DESCRIPTION:
The objective of this observational study is to assess the effectiveness and long-term clinical outcomes of various neoadjuvant immunotherapies in patients with non-small cell lung cancer (NSCLC), using the real-world data. The primary inquiries it seeks to address include:

* What is the optimal strategy for utilizing immune checkpoint inhibitors as neoadjuvant therapy?
* How can we identify specific patient subgroups that derive the greatest benefit from neoadjuvant immunotherapy? Participants will undergo neoadjuvant immunotherapy, and the study will meticulously analyze real-world data to provide insights into these pivotal questions, contributing to the refinement of treatment strategies and patient care in NSCLC management.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of non-small cell lung cancer (Stage I-IV, International Association for the Study of Lung Cancer staging eighth edition)
2. Patients who have previously undergone immune checkpoint inhibitors as the neoadjuvant treatment;
3. No previous history of malignant tumors and other malignant tumors at the same time, without any anti-tumor treatment;
4. Eastern Cooperative Oncology Group (ECOG) score 0-1, heart, lung, liver, brain and kidney function can tolerate surgery;
5. At least one measurable lesion (RECIST v1.1).

Exclusion Criteria:

1. Patients included in unblinded clinical trials or anti-tumor drug intervention.
2. Radiotherapy or systemic therapy were used for NSCLC patients before the surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients receiving neoadjuvant immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | Within 15 days after surgery
  defined as 0% of viable tumor cells in primary tumor and lymph nodes
Disease-free survival (DFS) | DFS was defined as the time from surgery to the date of disease recurrence or death (by any cause in the absence of recurrence), up to about 10 years.
  Defined as the time from the date of randomization until the date of disease recurrence or death (by any cause in the absence of recurrence).

SECONDARY OUTCOMES:
Overall survival (OS) | From date of surgery until date of death due to any cause, up to approximately 10 years.
  OS is defined as the time from surgery time until death from any cause.
Event-free survival (EFS) | EFS was defined as time from first dose date to disease progression, death, or discontinuation of treatment, up to approximately 10 years.
  EFS was defined as time from study inclusion (first dose date) to disease progression, death, or discontinuation of treatment.
Major Pathological Response (MPR) | Within 15 days after surgery
  defined as ≤10% of viable tumor cells
Relapse Patterns | Within 10 years after surgery
  Relapse was defined as disease recurrence at any site.

CONTACTS AND LOCATIONS:
Overall Officials: Shugeng Gao, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Shugeng Gao, Beijing, Beijing Municipality, China